CLINICAL TRIAL: NCT02711306
Title: Office of Human Research, Taipei Medical University
Brief Title: Effects of Konjac Glucomannan Noodle Intervention in Subjects With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 201209019
Record Dates: First submitted 2016-01-06; First posted 2016-03-17 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2013-03

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GMN Diet (Experimental): In the glucomannan noodle (GMN) diet, the participants received two servings (400 g) of GMN every day to replace their daily carbohydrate intake for 4 weeks, with each serving of glucomannan noodles weighing up to 200 g with 2 g of glucomannan.
  Interventions: Dietary Supplement: Glucomannan noodle; Dietary Supplement: Placebo noodle
- PN Diet (Placebo Comparator): In the placebo noodle (PN) diet, the participants received the participants received the same amount of noodles without glucomannan.
  Interventions: Dietary Supplement: Glucomannan noodle; Dietary Supplement: Placebo noodle

INTERVENTIONS:
Dietary Supplement: Glucomannan noodle — The participants received two servings (400 g) of GMN every day to replace their daily carbohydrate intake for 4 weeks.
Dietary Supplement: Placebo noodle — In the placebo noodle diet, the participants received the same amount of noodles without glucomannan for 4 weeks.

SUMMARY:
Metabolic syndrome (MS) is a complex disease with a cluster of risk factors and clinical features, which includes central or abdominal obesity, atherogenic dyslipidemia, impaired glucose regulation, hyperinsulinemia, high blood pressure, and concomitance of pro-inflammatory cytokine and insulin resistance. Glucomannan (GM) is a water-soluble dietary fiber derived from the root of Amorphophallus konjac that can improve blood sugar, blood fat concentration, and weight management, and has other health benefits.The purposes of this study are going to investigate the effects of KGM noodle (KGN) as stable food to MS and diabetic patients.

DETAILED DESCRIPTION:
The KGN diet was composed of well-cooked noodle with 2 g of KGM in a dosage of 200 g/piece twice daily to substitute the daily carbohydrate for 4 weeks, with a 2-week washout period between alternative diets. All 33 subjects received two servings of either GMNs or PNs (400 g) per day, which replaced the main carbohydrate in two daily meals for 4 weeks. After a 2-week washout period, the subjects received the other type of noodle for 4 weeks. The body weight, BMI, waist circumference, fasting blood glucose and lipid profile, as well as serum vitamin A, E, β-carotene and high sensitivity C-reactive protein (hs-CPR) were measured by HPCL.

ELIGIBILITY:
Inclusion Criteria: Adults with metabolic syndrome

Subjects were considered to have metabolic syndrome if subjects had 3 of the following 5 characteristics:

1. Abdominal obesity (waist circumference >= 90 cm in men and >= 80 cm in women)
2. Impaired fasting glucose ( >= 5.6 mmol/L)
3. Hypertriglyceridemia ( >= 1.7 mmol/L)
4. Low HDL-C (< 1.0 mmol/L in men and < 1.3 mmol/L in women)
5. Increased blood pressure (SBP >= 130 mmHg and DBP >= 85 mmHg).

Exclusion Criteria:

1. Liver and renal diseases
2. Undergoing statin therapy
3. Pregnancy women
4. Taking antioxidant vitamins supplements

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Han Lin, MS, Principal Investigator — Office of Human Research, Taipei Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sood N, Baker WL, Coleman CI. Effect of glucomannan on plasma lipid and glucose concentrations, body weight, and blood pressure: systematic review and meta-analysis. Am J Clin Nutr. 2008 Oct;88(4):1167-75. doi: 10.1093/ajcn/88.4.1167. PMID 18842808

RESULTS

PARTICIPANT FLOW:
Groups:
- First GMN Then PN: "First Intervention (4 weeks, GMN)", "Washout (2 weeks)" and "Second Intervention (4 weeks, PN)"
- First PN Then GMN: "First Intervention (4 weeks, PN)", "Washout (2 weeks)" and "Second Intervention (4 weeks, GMN)"
Period: Overall Study
Arm/Group | First GMN Then PN | First PN Then GMN
Started | 18 | 18
Completed | 16 | 16
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | First GMN Then PN | First PN Then GMN | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.75 (4.96) | 49.82 (12.59) | 50.79 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: Body weight by weighting scale (kilogram). Lower scores mean a better outcome in subjects.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | GMN Diet | PN Diet
Number analyzed (Participants) | 32 | 32
kg
  Baseline | 75.2 (10.86) | 74.97 (11.44)
  End | 74.41 (10.49) | 74.39 (11.27)

2. Secondary Outcome: Waist Circumference
Description: Body waist by tape in centimeter
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | GMN Diet | PN Diet
Number analyzed (Participants) | 32 | 32
cm
  Baseline | 92.03 (6.69) | 91.14 (7.26)
  End | 90.17 (6.8) | 90.15 (7.11)

3. Secondary Outcome: Glycemic Index
Description: HbA1c (glycated hemoglobin) analysis
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | GMN Diet | PN Diet
Number analyzed (Participants) | 32 | 32
percentage
  Baseline | 7.28 (1.65) | 7.21 (1.69)
  End | 7.08 (1.54) | 7.12 (1.6)

4. Secondary Outcome: Lipid Index
Description: LDL-C (low density lipoprotein cholesterol) analysis
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | GMN Diet | PN Diet
Number analyzed (Participants) | 32 | 32
mg/dL
  Baseline | 133.86 (32.54) | 135.39 (28.02)
  End | 137.24 (33.99) | 130.53 (33.63)

ADVERSE EVENTS:
Time Frame: The adverse event data were collected from the participants during intervention and assessed after 6 months.
Description: Adverse events were reported in real time, as they occurred (if any) by a physician who saw the subjects each day. As this was a dietary analysis/no pharmacological intervention, no adverse events were expected.
Groups:
- GMN Diet: The 100 g GMN noodle contains 1 g of konjac glucomannan powder. Participants approximately consumed 2 g GMN per day in 200 g of noodle. The intervention period was 4 weeks long. Meanwhile, the participants remained their usual eating habits except consuming any probiotics or prebiotics.
- PN Diet: Isocaloric noodle with no konjac glucomannan powder in placebo comparator. The PN-participants daily consumed placebo noodle without any added GMN (approximately 200 g noodle per day). The intervention period was 4 weeks long. Meanwhile, the participants will remain their usual eating habits except consuming any probiotics or prebiotics.
Arm/Group | GMN Diet | PN Diet
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No